CLINICAL TRIAL: NCT02160691
Title: Examining the Efficacy of the Anxiety Meter for Recognition and Management of Anxiety Signs in Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Azadeh Kushki, Scientist, Holland Bloorview Kids Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANXMT_RCT1
Record Dates: First submitted 2014-06-05; First posted 2014-06-11 (Estimated); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anxiety Meter (Experimental): The Anxiety Meter (experimental) group will receive a real-time display of physiological arousal on the Anxiety Meter during the intervention period in visit #4.
  Interventions: Device: Anxiety Meter
- No Anxiety Meter (No Intervention): The control group will have the Anxiety Meter during the intervention period, but the marker will not move.

INTERVENTIONS:
Device: Anxiety Meter — This is a new device developed to measure changes in heart rate and translate these into a visual display of arousal level in children with autism spectrum disorder.
  Arms: Anxiety Meter

SUMMARY:
The purpose of the study is to determine if a new device, called the Anxiety Meter, improves recognition and management of psychological arousal associated with anxiety in children with ASD.

DETAILED DESCRIPTION:
Anxiety is a prevalent, persistent, and disabling co-morbidity of autism spectrum disorder (ASD). In addition to its profound negative impact on physical and mental health, anxiety interacts with the core deficits of ASD to exacerbate symptomatology and increase functional impairment. Anxiety treatments efficacious in non-ASD children (e.g., Cognitive-Behavioural Therapy (CBT)) often have reduced potency and limited applicability in the ASD population due to impairments in cognitive ability, communication, emotional awareness, and introspection. Despite the urgency to treat co-morbid anxiety in ASD, there is limited evidence supporting treatment programs in higher-functioning individuals, and no evidence for those who are lower-functioning. In light of the urgent need for treatment of co-morbid anxiety in ASD and the paucity of evidence in this area, the investigators propose a study to establish early evidence on a technology-supported treatment of anxiety in children with ASD. This approach aims to reduce ASD-related barriers to treatment (e.g., deficits in emotional awareness and introspection) by providing children with a visual, real time display of their arousal level.

The proposed treatment focuses on the physiological arousal associated with anxiety. In particular, the investigators propose to use a physiological indicator of anxiety that can objectively measure and promote awareness of physiological arousal. To this end, the investigators have developed the Anxiety Meter, a device that measures arousal-related increases in heart rate using non-invasive wearable sensors and translates these to a visual display of the child's arousal level on a tablet computer. The investigators research questions are:

1. Primary: Does the Anxiety Meter improve awareness and management of physiological arousal induced by anxiogenic stimuli in a controlled setting? Hypothesis: The Anxiety Meter will improve awareness and management of symptoms because it promotes awareness of arousal - a skill which is impaired in ASD.
2. Secondary: What demographic and cognitive and behavioural variables predict response to the Anxiety Meter? Hypothesis: Age, IQ, sex, and severity of anxiety symptoms at baseline will affect treatment response.

To investigate the above questions, the investigators propose a randomized controlled trial comparing the Anxiety Meter to a control condition in children with ASD. Both the treatment and control groups will be taught a relaxation technique (three training sessions) and will be asked to apply the technique in a controlled anxiety-inducing task (one testing session). During the testing session, participants will be seated in front of a computer screen and will complete five tasks:

1. Baseline (30 minutes): After completing the STAI, participants will watch an animated movie clip. This task has been used successfully as a "baseline activity" in our previous studies in the target population.
2. Anxiety condition 1 (3 minutes): In this task, participants will be given 3 minutes to prepare a 3-minute talk. They will be told that the talk will be delivered to an audience of 3 strangers.
3. Intervention (2 minutes): Both groups will use this time to reflect on their anxiety level and apply the relaxation technique if they feel anxious. The treatment group will receive a real-time display of physiological arousal on the Anxiety Meter, whereas the control group will not receive feedback from the device. Our previous studies indicate that five minutes is sufficient for the heart rate to return to baseline. Both groups will complete the STAI (attached) as a report of their anxiety levels before and after the task.
4. Anxiety condition 2 (3 minutes): Participants will deliver a 3-minute talk to an audience of 3 strangers.
5. Return-to-baseline (15 minutes): Participants will watch an animated movie clip.

ELIGIBILITY:
Inclusion Criteria:

1. Children 8-18 years of age.
2. Primary diagnosis of autism spectrum disorder according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5).
3. Full-scale intelligence quotient (IQ) >50.
4. Must be able to complete tasks and the relaxation technique. A participant will be deemed able to do the public speaking task if he/she is able to complete Modules 3 or 4 of the Autism Diagnostic Observation Schedule (ADOS) protocol.
5. Must show physiological arousal in response to anxiety-inducing stimulus (minimum 2 beats/minute increase in heart rate).

Exclusion Criteria:

1. Started other treatments within four weeks at the time of the study.
2. Completed Cognitive Behavioural Therapy in the past.
3. Using beta-blockers.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Proportion of responders | Week 4
  We hypothesize that the proposed intervention will improve the recognition of arousal signs. To examine this hypothesis, our primary outcome measure is the proportion of participants initiating diaphragmatic breathing during the intervention period.

SECONDARY OUTCOMES:
Change in heart rate | Week 4
  We also hypothesis that the intervention will improving the potency of the relaxation technique through enhancing the participant's ability to sustain the breathing until relaxation is achieved. To examine this hypothesis, we will examine the difference in average heart rate between the anxiety (public speaking preparation) and post-intervention periods (public speaking delivery). Heart rate will be obtained from an electrocardiogram (ECG) sensor from Shimmer Research.
Change in self-reported anxiety level | Week 4
  To further examine the hypothesis that the intervention improves symptom management, change in self-reported anxiety level measured by the State-Trait Anxiety Inventory will be examined.The change will be measured between reports obtained before and after the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Azadeh Kushki, PhD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Nguyen J, Cardy RE, Anagnostou E, Brian J, Kushki A. Examining the effect of a wearable, anxiety detection technology on improving the awareness of anxiety signs in autism spectrum disorder: a pilot randomized controlled trial. Mol Autism. 2021 Nov 14;12(1):72. doi: 10.1186/s13229-021-00477-z. PMID 34775994